CLINICAL TRIAL: NCT02626624
Title: CarboClear Pedicle Screw System
Brief Title: Safety and Efficacy of the CarboClear Pedicle Screw System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CarboFix Orthopedics Ltd. (Industry)
Collaborators: CarboFix Orthopedics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARBOCLEAR P_CLD 2492_US
Record Dates: First submitted 2015-11-30; First posted 2015-12-10 (Estimated); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis, Grade 1
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- single arm (Experimental): CarboClear Pedicle Screw System
  Interventions: Device: Implantation of the CarboClear Pedicle Screw System

INTERVENTIONS:
Device: Implantation of the CarboClear Pedicle Screw System

SUMMARY:
The purpose of this trial is to demonstrate the safety and effectiveness of the CarboClear Pedicle Screw System, for skeletally mature DDD patients undergoing one level spinal fusion in combination with interbody fusion device, and requiring immediate, rigid, posterior spinal stabilization of the lumbar and/or sacral spine.

DETAILED DESCRIPTION:
A prospective, multi-center, confirmatory, single arm, study. Results of the study will be compared to data from the literature.

The CarboClear Pedicle Screw System is designed for use with intervertebral body fusion device and with autogenous and/or allogenic bone graft comprised of cancellous and/or corticocancellous bone graft, using PLIF or TLIF.

A total of 55 subjects will participate in the study, with up to 25 patients recruited at sites in Israel and at least 30 patients will be enrolled in US sites.

Follow-ups: Radiographic (AP, lateral and flexion/extension X-Rays) and clinical evaluations.

Follow-up sessions at 6 weeks, 3 months, 6 months, 12 months, and 24 months postoperatively, and then annually, until the last patient has completed 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has degenerative disc disease (DDD) at one level, from L2 to S1 vertebrae, with up to Grade I spondylolisthesis.

   DDD is defined as back pain and/or radicular leg pain with degeneration of the disc confirmed by patient history, radiographic studies, and physical examination, with one or more of the following factors (as measured radiographically, either by CT, MRI or plain film, myelography, discography, etc.):
   * osteophyte formation of facet joints or vertebral endplates;
   * decreased disc height, on average by > 2 mm;
   * scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule;
   * herniated nucleus pulposus;
   * facet joint degeneration/changes;
   * vacuum phenomenon.
2. Subject is candidate for single level intervertebral fusion, with or without posterolateral fusion, with implantation of intervertebral body fusion device and supplemental fixation.
3. Subject age is between 21 - 72 years, and subject is skeletally mature.
4. Pre-operative low back and/or leg/s pain (debilitating pain that causes a significant disturbance of the routine daily physical activities) ≥ 40 mm on a 100 mm Visual Analogue Scale (VAS).
5. Pre-operative Oswestry Disability Index (ODI) score ≥ 40 percentage-point, indicating at least moderate disability (interpreted as moderate/severe disability).
6. Low back and/or leg/s pain is unresponsive to prior non-surgical management for a minimum of six months. Non-operative treatment includes pain medication, physical therapy and/or injections.
7. Patient must understand and sign the informed consent.
8. Patient is willing and able to meet the proposed follow-up schedule including return to follow-up visits and complete necessary study paperwork.
9. Patient is willing and able to follow the postoperative management program.

Exclusion Criteria:

1. Previous fusion or fusion attempts, including anterior fusion or posterolateral fusion, at the index level.
2. Previous fusion or fusion attempts at the adjacent levels.
3. Prior decompression procedures that include removal of soft and bone tissue at the index or adjacent levels.
4. Patient is not skeletally mature.
5. Degenerative spondylolisthesis greater than Grade I.
6. Spinal instability at the index level with ≥ 3 mm translation and/or ≥ 5 degrees angulation. Determination of instability will be assessed using flexion/extension lateral view radiographs.
7. Isthmic spondylolisthesis.
8. Radiographically confirmed moderate or severe spinal stenosis with associated neurogenic claudication. Radiographically confirmed moderate/severe stenosis is defined as reduction of ˃50% of central and/or foraminal canal diameter compared to the adjacent uninvolved levels. Neurogenic claudication is leg, groin or buttock pain and/or numbness that worsens with walking or erect posture and is relieved with flexion of the spine.
9. Systemic infection or infection at the site of surgery.
10. Metabolic bone disease, such as osteopenia, osteoporosis, and osteomalacia. A screening Questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a DEXA bone mineral density measurement. If DEXA is required, exclusion will be defined as measured T-score less than or equal to -2.5 (WHO definition).
11. History of Paget's disease or other bone pathologies, whether acquired or congenital, including renal osteodystrophy, untreated or uncontrolled hyperthyrodism, hypothyroidism, hyperparathyroidism, Ehrlers-Danlos-syndrome, osteogenesis imperfecta, achondroplasia, tuberculosis.
12. Personal and/or familial history NF2, and/or spinal tumor.
13. Ankylosing spondylitis.
14. Diffuse idiopathic skeletal hyperostosis (DISH) syndrome.
15. Active hepatitis (viral or serum) or HIV positive, renal failure, systemic lupus erythematosus, or any other significant medical conditions which would substantially increase the risk of surgery.
16. Immune deficiency disease.
17. Patient is receiving immunosuppressive or long-term steroid therapy.
18. Active malignancy or other significant medical comorbidities.
19. All concomitant diseases that can jeopardize the functioning and success of the patient.
20. Allergy to any component of the investigational device, including carbon fiber-reinforced polyetheretherketone (CFR-PEEK), titanium, and tantalum.
21. Pregnancy, or female subject interested in become pregnant during the duration of the study.
22. Current chemical dependency (e.g., drug and/or alcohol abuse, according to DSM-V definition), as well as those with a history of such abuse.
23. Uncontrolled depression, psychosis, or other symptoms of a mental disorder that, in the investigator's opinion, likely would make the subject unable to comply with the study procedures and could affect the study outcome.
24. Treatment with drugs that may interfere with bone metabolism, such as glucocorticosteroids, calcitonin, bisphosphonates, bone therapeutic doses of fluoride, bone therapeutic doses of vitamin D or vitamin D metabolites, and treatment by chemotherapy.
25. Morbid obesity (BMI ≥ 40).
26. Current smokers (including 3 months prior to surgery).
27. Scoliosis, Cobb angle greater than 11°.
28. Vertebral fractures.
29. Severe muscular, neural or vascular diseases that endanger the spinal column.
30. Missing bone structures, due to severely deformed anatomy or congenital anomalies, which make good anchorage of the implant impossible.
31. Paralysis.
32. Current use of other investigational drug or device.
33. The patient is involved in a worker's compensation case or spine-related litigation.
34. The patient is a prisoner.

Ages: 21 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-12-27 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Brooklyn Hospital, Brooklyn, New York
  - Crystal Clinic Orthopaedic Center, Akron, Ohio
  - St. David's Round Rock Medical Center, Austin, Texas
- Israel (3):
  - Herzliya Medical Center, Herzliya
  - Meir Medical Center, Kfar Saba
  - Assuta Medical Center - Israel Spine Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The single arm study was approved for a total of 55 subjects, and was conducted at 5 US sites and 3 Israeli sites.
Pre-assignment Details: A one arm study (no assignment to groups)
Groups:
- CarboClear Pedicle Screw System (Single Arm Study): Patients with Degenerative Disc Disease (DDD) at one level (L2-S1), aged 21-71 years, who have failed to improve with conservative treatment with at least 6 months prior to enrolment.
  Implantation of the CarboClear Pedicle Screw System and interbody spinal fusion using an FDA cleared PEEK interbody fusion device (PLIF or TLIF approach); and posterolateral spinal fusion at the physician's discretion.
Period: Overall Study
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Started | 57 (Study was approved for 55 pts, and extended after approval to 57, to replace 2 pts who died prior to significant data collection [one pt, with cardiac history (underwent in the past bypass surgery and 3 stenting): operation was completed uneventful, and upon emergence form anesthesia had cardiac arrest. 2nd pt: committed suicide 7 months postop.; pt had no neurological impairment/complication]. Their death was determined by the independent Clinical Event Committee as not related to the device.)
Completed | 47 (Four patients did not stop smoking, in contrary to the eligibility criteria, and were determined to be major protocol violation and excluded from the analysis.)
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 4
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 57
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 55.16 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55
  African | 2
Region of Enrollment [Number; unit: participants]
  United States | 31
  Israel | 26
Indications [Count of Participants; unit: Participants] — DDD = degenerative disc disease Mild spinal stenosis = reduction of up to 50% of central and/or foraminal canal diameter compared to the adjacent uninvolved levels
  Participants
    DDD + Spondylolisthesis up to Grade I + Mild Stenosis (< 50%) | 53
    DDD + Spondylolisthesis up to Grade I | 1
    DDD + Mild Stenosis (< 50%) | 2
    DDD | 1
Pain using Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — Patient self-assessed VAS questionnaire was used for measuring lower back pain and both legs pain. Each VAS score is determined from measurements of responses to pain question for each location (i.e., low back, right leg, and left leg), provided on a 100 mm scale. The anchor points are "No Pain" (0 mm) and "Severe Pain" (100 mm). Population: Mean VAS is calculated for subjects with preoperative VAS pain ≥ 40 mm on a 100 mm VAS (which is regarded as debilitating pain that causes a significant disturbance of the routine daily physical activities).
  units on a scale
    Lower Back Pain (VAS) | 81.83 (17.60)
    Right Leg Pain (VAS) | 61.80 (34.97)
    Left Leg Pain (VAS) | 56.32 (37.45)
Function using Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — The ODI questionnaire is based on patient's responses to 10 questions, each has 6 possible answers. The responses to each question ranges from 0-5 points. A lower numeric score represents a lower pain and disability status regarding that variable. A total ODI score is the sum of the scores of the individual questions, divided by the maximum possible total score (50). ODI score is presented in a range of 0%-100%, with a lower percentage indicating less pain and disability.
  units on a scale | 57.71 (12.14)

OUTCOME MEASURES:

1. Primary Outcome: Fusion: Evaluated Radiographically (by AP, Lateral and Flexion/Extension X-Rays) by Independent Radiographic Core Lab.
Description: Fusion was assessed at follow-up visits, starting at 6 months post operation.
  Fusion is defined as:
  1. Angular motion ˂ 3º; AND
  2. Translational motion ˂ 3 mm; AND
  3. Presence of continuous bridging bone between the involved motion segment, i.e.:
     * Presence of interbody (between endplates) bridging bone and absence of radiolucency > 50%; OR
     * Presence of right posterolateral bridging bone; OR
     * Presence of left posterolateral bridging bone.
Time Frame: 24 months
Population: 24-month radiographic data is available for 49 patients (for patients that attended the 24-month visit, or for non-attendees for whom data is available from earlier visits (e.g., where fusion was confirmed).
Measure: Count of Participants; unit: Participants
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 49
Participants | 42

2. Primary Outcome: Pain (Low Back and/or Leg/s): Assessed Based on Visual Analogue Scale (VAS) Patient Questionnaire
Description: Pain was assessed using the Visual Analogue Scale (VAS) preoperatively and at follow-up visits.
  The scale ranges from 0 mm ("No Pain") to 100 mm ("Severe Pain"). Patients were instructed to draw a single line across the scale at the point that best described their level of pain.
  Pain improvement was evaluated at each location (i.e., low back, right leg, and left leg) and was defined as a reduction of at least 20 mm on a 100 mm VAS from baseline level at 24 months.
  Eligible patients experienced preoperative low back and/or leg pain (debilitating pain that significantly disrupted daily physical activities) with a VAS score of ≥40 mm.
Time Frame: 24 months
Population: VAS pain data is available at 24 months for 45 patients who attended 24-month visit and for whom VAS assessment is available.
  Analysis is presented for patients with preoperative pain VAS score ≥40 (in accordance with the clinical investigational plan).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 45
score on a scale
  Pain Improvement (VAS) - Low Back: number analyzed (Participants) | 44
  Pain Improvement (VAS) - Low Back | 58.52 (31.89)
  Pain Improvement (VAS) - Right Leg: number analyzed (Participants) | 32
  Pain Improvement (VAS) - Right Leg | 58.11 (35.46)
  Pain Improvement (VAS) - Left Leg: number analyzed (Participants) | 28
  Pain Improvement (VAS) - Left Leg | 59.06 (32.99)

3. Primary Outcome: Function: Assessed by Oswestry Disability Index (ODI) Patient Questionnaire
Description: The Oswestry Disability Index (ODI) is a patient-reported questionnaire administered preoperatively and at follow-up visits. The ODI consists of ten questions focusing on pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. Each question has six possible responses.
  The response scale ranges from 0 to 5 points, with a lower score indicating better function and lower pain (0 points for full functionality with no or minimal pain; 5 points for inability to perform the function due to pain). The total ODI score is calculated by summing the individual question scores and dividing the total by the maximum possible score (50 if all questions are answered), yielding a percentage. ODI scores range from 0% to 100%, with lower percentages indicating reduced pain and disability.
  The functional outcome measure was defined as an improvement of at least 15 points from baseline at 24 months.
Time Frame: 24 months
Population: Function (ODI) data is available at 24 months for 45 patients who attended 24-month visit and for whom function assessment is available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 45
score on a scale | 34.39 (21.43)

4. Primary Outcome: Safety: Neurological Deterioration, Device Related Serious Adverse Events, Additional Surgical Intervention at Index Level.
Description: 1. Worsening in neurological status (motor, sensory, reflex, straight leg raising, and tenderness assessments) and no new permanent neurological deficits present for at least 2 successive visits at or beyond 6 months (out to 24 months);
  2. Device-related serious adverse events (SAEs) through 24 months;
  3. Subsequent surgical interventions at the index level through 24 months.
Time Frame: Throughout the study until 24 months
Population: All subjects that completed the study the study
Measure: Count of Participants; unit: Participants
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 55
Participants
  Neurological deterioration | 3
  Device related serious adverse events | 0
  Subsequent surgical interventions at the index level | 4

5. Secondary Outcome: Subject's Overall Well-Being: Assessed by 12-Item Short Form Health Survey (SF-12) Patient Questionnaire
Description: Subject's overall well-being (quality of life) was assessed preoperatively and at follow-up visits, using the 12-Item Short Form Health Survey (SF-12), which is a multipurpose short-form quality of life instrument with 12 questions selected from the SF-36 Health Survey. SF-12 questionnaire is designed to measure general health status from the patient's point of view. Results are expressed in terms of two meta-scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The PCS Score is a composite of the Physical Functioning, Role Functioning, Bodily Pain and General Health Scales within the SF-12 instrument. The MCS is a composite of the Vitality, Social Functioning, Role-Emotional and Mental Health Scales within the SF-12 instrument. The SF-12 is a normative based instrument. PCS and MCS are computed using the rating on 12 questions from 0 to 100, where a 0 score indicates the lowest level of health and 100 indicates the highest level.
Time Frame: 24 months
Population: Out of the patients attended the 24-month visit, 43 patients had SF-12 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 43
score on a scale
  SF-12 PCS Change | 14.50 (14.45)
  SF-12 MCS Change | 10.45 (13.90)

6. Secondary Outcome: Patient Satisfaction: Assessed Based on VAS Patient Questionnaire.
Description: Satisfaction was assessed at postoperative follow-up visits including at 24-month visit, using a 100 mm VAS (the anchor points are "Completely Not Satisfied" (0 mm) and "Completely Satisfied" (100 mm)).
  Pain was assessed using the Visual Analogue Scale (VAS) preoperatively and at follow-up visits.
  The scale ranges from 0 mm ("No Pain") to 100 mm ("Severe Pain"). Patients were instructed to draw a single line across the scale at the point that best described their level of pain.
  Pain improvement was evaluated at each location (i.e., low back, right leg, and left leg) and was defined as a reduction of at least 20 mm on a 100 mm VAS from baseline level at 24 months.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 45
score on a scale | 81.19 (32.20)

7. Secondary Outcome: Operation Time [Min]
Description: Operation time (skin-to-skin) was recorded for each subject.
Time Frame: During operation (skin-to-skin)
Population: All 55 patients that participated in the study
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 55
minutes | 135.20 (73.38)

8. Secondary Outcome: Blood Loss During Operation [ml]
Description: The volume of blood loss during operation was recorded for each subject.
Time Frame: During operation (skin to skin)
Population: All 55 patients that participated in the study
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
Number analyzed (Participants) | 55
milliliter | 212.64 (127.90)

ADVERSE EVENTS:
Time Frame: Evaluation of complications/adverse events was conducted at each follow-up session, as well as throughout the study (within 24 months).
Description: All adverse events (AEs), including non-serious AEs, non-device related, and anticipated AEs, were assessed by an independent Clinical Events Committee (CEC). AEs and serious adverse events (SAEs) were defined in accordance with the definition of ISO 14155.
Arm/Group | CarboClear Pedicle Screw System (Single Arm Study)
All-Cause Mortality (participants affected / at risk) | 2/57
Serious Adverse Events (participants affected / at risk) | 7/57
Other Adverse Events (participants affected / at risk) | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CarboClear Pedicle Screw System (Single Arm Study) (N=57)
Additional Surgery at index level (Surgical and medical procedures) | 4 (4) — Two additional surgeries due to hematoma/seroma; one replacement of a misplaced screw a day after surgery; and one replacement of the device 3 months post-operation due to intractable back pain (CEC noted that indicate screws were relatively short).
Additional surgery at non-index level (Surgical and medical procedures) | 2 (2) — One patient had additional surgery a few days post-operation to remove disc fragment below index level; another patient had operation to treat adjacent level after about 2 years.
Deep vein thrombosis (Vascular disorders) | 1 (1) — One patient had DVT 2 weeks post-op., developed to pulmonary emboli and right heart strain. Resolved after a few days.

LIMITATIONS AND CAVEATS:
This IDE study encountered a challenging follow-up schedule due to the COVID-19 pandemic. In particular, for several subjects, the 24-month visit occurred during the pandemic period, and was the cause for not attending this visit. On top of quarantine and limitations posed by authorities, a few subjects refused to arrive to hospital during that period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02626624/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02626624/ICF_001.pdf